CLINICAL TRIAL: NCT04973748
Title: Open-label Conditioning Therapy for Peri-operative Pain Management in Head and Neck Cancer Patients
Brief Title: Conditioned Open-label Placebo (COLP) for Peri-operative Pain Management in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00276225
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Opioid Use
Keywords: open label placebo; opioid; postoperative analgesia; placebo; head and neck cancer
MeSH Terms: conditions — Pain, Postoperative; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): Standard pain regimen with scheduled acetaminophen and ibuprofen, oxycodone as needed for moderate-to-severe pain, and intravenous hydromorphone as needed for breakthrough pain.
  Surveys about pain levels, opioid consumption, side effects of opioids, understanding of placebo effect and symptoms of depression.
  Interventions: Behavioral: Surveys about pain, opioid use and depression symptoms
- Conditioned open-label placebo (COLP) (Experimental): Standard pain regimen with scheduled acetaminophen and ibuprofen, oxycodone as needed for moderate-to-severe pain, and intravenous hydromorphone as needed for breakthrough pain.
  Conditioning (i.e. exposure to clove oil scent) with each dose of oxycodone medication on post-operative day (POD) 1-5.
  Scheduled placebo oxycodone medication paired with conditioning (i.e. exposure to clove oil scent) 3 times per day on POD 2-5.
  Surveys about pain levels, opioid consumption, side effects of opioids, understanding of placebo effect and symptoms of depression.
  Interventions: Behavioral: Conditioned open-label placebo (COLP); Behavioral: Surveys about pain, opioid use and depression symptoms

INTERVENTIONS:
Behavioral: Conditioned open-label placebo (COLP) — Placebo oxycodone will be formulated to have the same physical appearance as liquid oxycodone and will be dispensed by the inpatient pharmacy and administered by the nursing staff. At all times that oxycodone or placebo medication is administered on post-operative day (POD) 1-5, the patient will undergo conditioning via exposure to a clove oil scent:
  1. Conditioning (i.e. exposure to clove oil scent) with each dose of oxycodone medication on POD 1-5.
  2. Scheduled placebo oxycodone medication paired with conditioning (i.e. exposure to clove oil scent) 3 times per day on POD 2-5.
  Arms: Conditioned open-label placebo (COLP)
Behavioral: Surveys about pain, opioid use and depression symptoms — Surveys before surgery: Within 1 week prior to surgery, patients complete surveys about pain levels, opioid consumption, understanding of placebo effect and symptoms of depression.
  Surveys after surgery: Through 6-months after surgery, patients complete surveys about pain levels, opioid consumption, side effects of opioids and symptoms of depression.

SUMMARY:
The opioid epidemic is a considerable problem in the United States, and prescription opioids significantly contribute to the epidemic. Head and neck cancer (HNC) patients are inherently at increased risk for opioid dependence as surgical treatment can cause significant pain and up to 50% of patients also suffer from psychiatric comorbidities. Novel methods are needed to decrease opioid consumption following HNC surgeries to limit the risk of chronic opioid dependence in these patients. Conditioning therapy with placebo aims to elicit a classically conditioned response to an inactive medication through consistent pairing of the medication with a neutral stimulus (i.e. an odor) and has been shown to be effective for decreasing the amount of active drug require for certain clinical responses, including for acute pain. However, studies have not been completed for the treatment of acute pain in the inpatient post-operative setting. The overall goal of this pilot study is to determine the feasibility and effectiveness of conditioned open-label placebo (COLP) as an adjunct for post-operative pain management in complex head and neck cancer patients. This randomized, controlled, open-label trial will specifically compare post-operative opioid consumption and pain scales between patients receiving multimodal analgesia along with conditioned open-label placebo (COLP group) to those receiving multimodal analgesia, alone (Treatment as usual group). Findings from this study will determine the efficacy of COLP as an innovative approach to decrease opioid consumption and improve pain control in head and neck cancer patients and will provide rationale for development of future large scale trials.

DETAILED DESCRIPTION:
Background:

The opioid epidemic is a considerable problem in the United States, with more than 5 million Americans currently affected by opioid-related substance use disorders. While prescription medications may be thought of as safe and controlled, many opioid-naïve patients report continuing to take prescription opioids for over one year after surgery, and the majority of heroin users report starting with abuse of prescription opioids. At the same time, prescription opioids have more than doubled from 2001-2013 and multiple studies in other surgical specialties suggest that patients receive opioids in excess of the patient's peri-operative pain needs Prior efforts to battle this epidemic have included the increased use of multimodal analgesia, policies to limit the amount of opioids able to be prescribed at one time, and databases to track prescribing habits across health care facilities. While these have had some success, there is significant room for improvement.

Head and neck cancer (HNC) patients represent a unique population in that surgical resection often leads to significant peri-operative pain and disfigurement. A high proportion, up to 50% of these patients also suffer from psychiatric comorbidities. These factors inherently increase the risk of opioid dependence and studies have shown that chronic opioid use following surgery for HNC is associated with decreased disease free survival. Novel methods are needed to minimize opioid risks in this patient population.

Conditioning therapy aims to elicit a classically conditioned, or Pavlovian, response through consistent pairing of a medication with a neutral stimulus (i.e. an odor). Treatment involves reinforcement with simultaneous presentation of a characteristic odor with each dose of active and inactive medication. Prior studies have shown efficacy of conditioning therapy paired with placebo medication to decrease the total dose of active medications required for a clinical response including opioids for pain following spinal cord injury, stimulants for attention deficit hyperactivity disorder, and corticosteroids for psoriasis. Many of these have been performed as "open-label" studies, where patients were aware of group assignment and were informed when each placebo treatment was given.

These results suggest that patients with HNC may also benefit from conditioned open-label placebos by reducing total opioid consumption required for adequate pain control in the peri-operative setting and providing an innovative intervention to potentially decrease the risk of opioid dependence in this patient population.

Primary Objective:

Determine if the addition conditioned open-label placebo (COLP) to standard multimodal analgesia decreases baseline opioid consumption from post-operative day (POD) 2 to 5 in comparison to standard multimodal analgesia alone in patients with head and neck cancer.

Rationale:

Patients with head and neck cancer will be enrolled in this randomized, controlled, open-label trial. All study participants will receive standard multimodal analgesia, including opioids, and will have daily opioid consumption and pain severity documented following surgery. Patients in the COLP group will additionally receive conditioning (i.e. exposure to clove oil) with each active oxycodone dose on POD 1-5 and a scheduled placebo oxycodone paired with conditioning (i.e. exposure to clove oil) 3 times per day on POD 2-5. The chance in baseline opioid consumption from POD 2 to 5 will be compared between groups.

Secondary Objectives:

Determine if the addition conditioned open-label placebo (COLP) to standard multimodal analgesia leads to a reduction in pain severity following surgery and persistent opioid use at 6-months following surgery in comparison to standard multimodal analgesia alone in patients with head and neck cancer.

Rationale:

Following surgery, patients complete daily surveys on pain severity. The investigators will compare these pain scales between COLP and TAU groups to determine if there is a difference in pain severity between treatment groups. The investigators will also analyze long-term effects of the intervention with COLP. After the second week following surgery, opioid consumption will continue to be recorded by nursing (if inpatient) or with patient reported surveys (after discharge) through 6 months after surgery. While COLP may have immediate effects on opioid consumption during therapy, the goal of this aim is to determine if short-term therapy can result in long-term changes in behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving pre-operative evaluation for head and neck cancer in the Otolaryngology - Head and Neck Surgery Department at Johns Hopkins Hospital
* Scheduled for surgery for resection of and/or reconstruction following resection of a head and neck tumor between November 15, 2022 - May 15, 2024, with expected inpatient admission of at least 5 days after surgery.
* Age 18 years or older
* Ability to comprehend and willingness to participate in open-label conditioning portion of study regardless of study group assignment
* Ability to participate in study for 1 week prior to surgery and 6 months following surgery at time of enrollment

Exclusion Criteria:

* Past medical history of substance use disorder
* Chronic pain (defined as pain lasting >3 months) or chronic opioid use (for >3 months).
* Contraindication to receiving acetaminophen, ibuprofen, oxycodone, or hydromorphone
* New gabapentin prescription started <2 weeks prior to surgery
* Psychosis, delirium or other significant cognitive impairment preventing participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Change in baseline daily morphine milligram equivalents (MME/day) | once after surgery up to 1 week
  Comparison of average daily MME on POD 5 to average daily MME on POD 2 between TAU and COLP groups.

SECONDARY OUTCOMES:
Change in Pain assessed by Visual Analogue Scale | daily after surgery up to 2 weeks, then weekly daily after surgery up to 1 month, then monthly daily after surgery up to 3 months, then once daily after surgery up to 6 months
  Measurement of subjective pain; 0 = no pain to 100 = most intense pain ever experienced.
Change in Pain as assessed by the Functional Pain Scale | daily after surgery up to 2 weeks, then weekly daily after surgery up to 1 month, then monthly daily after surgery up to 3 months, then once daily after surgery up to 6 months
  Subjective measurement of how pain affects activities of daily living; 0 = no pain to 10 = intolerable pain where the patient cannot do any activity (even speak) because of pain.
Change in Depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | weekly daily after surgery up to 1 month, then monthly daily after surgery up to 3 months, then once daily after surgery up to 6 months
  Objectifies degree of depression; 0-4: none/minimal, 5-9: mild, 10-14: moderate, 15-19: moderately severe, 20-27: severe
Change in Numerical Opioid Side Effects (NOSE) | daily after surgery up to 2 weeks, then weekly daily after surgery up to 1 month, then monthly daily after surgery up to 3 months, then once daily after surgery up to 6 months
  Subjective measurement of severity of side effects related to opioid use; 0 = not present to 10 = as bad as you can imagine.
Persistent opioid consumption at 6 months after surgery | once after surgery up to 6 months
  Proportion of patients with opioid consumption 6 months after surgery between TAU and COLP groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Fakhry, MD, Principal Investigator — JHU SOM Oto Head and Neck Surgery
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data (i.e. counts/averages), will be shared after appropriate request. Individual de-identified data will not be shared given small number of participants in this trial.

REFERENCES:
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Lydiatt WM, Moran J, Burke WJ. A review of depression in the head and neck cancer patient. Clin Adv Hematol Oncol. 2009 Jun;7(6):397-403. PMID 19606075
- [Background] Hill MV, Stucke RS, Billmeier SE, Kelly JL, Barth RJ Jr. Guideline for Discharge Opioid Prescriptions after Inpatient General Surgical Procedures. J Am Coll Surg. 2018 Jun;226(6):996-1003. doi: 10.1016/j.jamcollsurg.2017.10.012. Epub 2017 Nov 30. PMID 29198638
- [Background] Dang S, Duffy A, Li JC, Gandee Z, Rana T, Gunville B, Zhan T, Curry J, Luginbuhl A, Cottrill E, Cognetti D. Postoperative opioid-prescribing practices in otolaryngology: A multiphasic study. Laryngoscope. 2020 Mar;130(3):659-665. doi: 10.1002/lary.28101. Epub 2019 Jun 21. PMID 31225905
- [Background] Buchmann L, Conlee J, Hunt J, Agarwal J, White S. Psychosocial distress is prevalent in head and neck cancer patients. Laryngoscope. 2013 Jun;123(6):1424-9. doi: 10.1002/lary.23886. Epub 2013 Apr 1. PMID 23553220
- [Background] Chan JY, Lua LL, Starmer HH, Sun DQ, Rosenblatt ES, Gourin CG. The relationship between depressive symptoms and initial quality of life and function in head and neck cancer. Laryngoscope. 2011 Jun;121(6):1212-8. doi: 10.1002/lary.21788. Epub 2011 May 3. PMID 21541945
- [Background] Starr N, Oyler DR, Schadler A, Aouad RK. Chronic opioid use after laryngeal cancer treatment. Head Neck. 2021 Apr;43(4):1242-1251. doi: 10.1002/hed.26591. Epub 2020 Dec 28. PMID 33368718
- [Background] Pang J, Tringale KR, Tapia VJ, Moss WJ, May ME, Furnish T, Barnachea L, Brumund KT, Sacco AG, Weisman RA, Nguyen QT, Harris JP, Coffey CS, Califano JA 3rd. Chronic Opioid Use Following Surgery for Oral Cavity Cancer. JAMA Otolaryngol Head Neck Surg. 2017 Dec 1;143(12):1187-1194. doi: 10.1001/jamaoto.2017.0582. PMID 28445584
- [Background] Ader R, Mercurio MG, Walton J, James D, Davis M, Ojha V, Kimball AB, Fiorentino D. Conditioned pharmacotherapeutic effects: a preliminary study. Psychosom Med. 2010 Feb;72(2):192-7. doi: 10.1097/PSY.0b013e3181cbd38b. Epub 2009 Dec 22. PMID 20028830
- [Background] Morales-Quezada L, Mesia-Toledo I, Estudillo-Guerra A, O'Connor KC, Schneider JC, Sohn DJ, Crandell DM, Kaptchuk T, Zafonte R. Conditioning open-label placebo: a pilot pharmacobehavioral approach for opioid dose reduction and pain control. Pain Rep. 2020 Jul 20;5(4):e828. doi: 10.1097/PR9.0000000000000828. eCollection 2020 Jul-Aug. PMID 32766465
- [Background] Sandler AD, Bodfish JW. Open-label use of placebos in the treatment of ADHD: a pilot study. Child Care Health Dev. 2008 Jan;34(1):104-10. doi: 10.1111/j.1365-2214.2007.00797.x. PMID 18171451
- [Background] Shunmugasundaram C, Rutherford C, Butow PN, Sundaresan P, Dhillon HM. What are the optimal measures to identify anxiety and depression in people diagnosed with head and neck cancer (HNC): a systematic review. J Patient Rep Outcomes. 2020 Apr 23;4(1):26. doi: 10.1186/s41687-020-00189-7. PMID 32328839
- [Background] Gloth FM 3rd, Scheve AA, Stober CV, Chow S, Prosser J. The Functional Pain Scale: reliability, validity, and responsiveness in an elderly population. J Am Med Dir Assoc. 2001 May-Jun;2(3):110-4. PMID 12812581
- [Background] Arnstein P, Gentile D, Wilson M. Validating the Functional Pain Scale for Hospitalized Adults. Pain Manag Nurs. 2019 Oct;20(5):418-424. doi: 10.1016/j.pmn.2019.03.006. Epub 2019 May 14. PMID 31101560
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928
- [Background] Cometto-Muniz JE, Cain WS, Abraham MH. Determinants for nasal trigeminal detection of volatile organic compounds. Chem Senses. 2005 Oct;30(8):627-42. doi: 10.1093/chemse/bji056. Epub 2005 Sep 1. PMID 16141291
- [Derived] Trakimas DR, Colloca L, Fakhry C, Tan M, Khan Z, Vosler PS. Study protocol: randomised controlled trial of conditioned open-label placebo (COLP) for perioperative pain management in patients with head and neck cancer. BMJ Open. 2023 Jul 7;13(7):e069785. doi: 10.1136/bmjopen-2022-069785. PMID 37419646